CLINICAL TRIAL: NCT02993276
Title: Protect Neuro - Prospective Cohort Evaluation of NEUROCAP® In the Treatment of Symptomatic Neuroma
Brief Title: Evaluation of NEUROCAP® In the Treatment of Symptomatic Neuroma
Status: Completed | Type: Observational
Sponsor: Polyganics BV (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-02
Record Dates: First submitted 2016-12-08; First posted 2016-12-15 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2019-09

CONDITIONS: Neuroma
MeSH Terms: conditions — Neuroma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Treatment Group: All subjects receiving the Neurocap® device when surgically treated for their symptomatic peripheral end-neuroma.
  Interventions: Device: Neurocap®

INTERVENTIONS:
Device: Neurocap® — NEUROCAP®, a bioresorbable nerve capping device based upon the NEUROLAC® nerve guide, is indicated to protect a peripheral nerve end and to separate the nerve from surrounding environment to reduce the development of a symptomatic neuroma.

SUMMARY:
PROSPECTIVE COHORT EVALUATION OF NEUROCAP® In the Treatment of symptomatic Neuroma (PROTECT Neuro)

This post-market surveillance study is conducted to provide post market surveillance information regarding long-term performance and ease of use of the Polyganics nerve capping device (NEUROCAP®) for reduction of the development of peripheral symptomatic end-neuroma.

DETAILED DESCRIPTION:
1. Device description NEUROCAP®, a bioresorbable nerve capping device based upon the NEUROLAC® nerve guide, is indicated to protect a peripheral nerve end and to separate the nerve from surrounding environment to reduce the development of a symptomatic neuroma. NEUROCAP® is composed of the same biocompatible, bioresorbable copolyester composing the NEUROLAC® nerve guide, Poly(68/32[15/85 D/L] Lactide-Ԑ-Caprolactone) (PLCL).
2. Objective This post-market surveillance study is conducted to provide post market surveillance information regarding long-term performance and ease of use of the Polyganics nerve capping device (NEUROCAP®) for reduction of the development of peripheral symptomatic end-neuroma.
3. Study design This post-market surveillance study consists of a cohort study to provide post market surveillance information regarding long-term performance and ease of use of the NEUROCAP® for reduction of the development of peripheral symptomatic end-neuroma in the upper and lower extremity. Sub analyses will be performed regarding demographics and medical background.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are able to provide a written informed consent prior to participating in the clinical investigation.
2. Subjects who are able to comply with the follow-up or other requirements.
3. Subjects who are ≥ 18 years old.
4. Subjects with a diagnosis of peripheral symptomatic (end-) neuroma in the upper limb.
5. Subjects with a positive Tinel's sign.
6. Symptomatic neuroma confirmed by pain relief following a 10min ± 2min nerve block with Xylocaine (Lidocaine) - Pain relief defined as minimally 50% reduction in VAS questionnaire score.
7. Subjects that are indicated for surgery to treat symptomatic neuroma.

Exclusion Criteria:

1. Subjects who do not complete the informed consent.
2. Subjects who are not willing to follow post-surgery protocols (e.g. avoiding pressure on the implant zone or immobilization).
3. Subjects who are unable to comply with the follow-up or other requirements and/or have a life expectancy of less than 24 months.
4. Subjects with congenital neuropathy.
5. Insufficient amount of soft tissue to cover the investigational device, as assessed by the surgeon. Use of the device over a joint is advised against.
6. Subjects who have had historical radiotherapy in the area of the (end-) neuroma.
7. Subjects who have a known allergy to anesthetic agent or bioresorbable copolyester Poly(68/32[15/85 D/L] Lactide-ε-Caprolactone) (PLCL).
8. Proximal nerve end > 8mm.
9. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Peripheral symptomatic end-neuroma patients indicated for surgical treatment of the neuroma.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) for Pain | 2 years
  Subjective pain score as indicated by the patient on a scale of 1-100.

SECONDARY OUTCOMES:
Recurrence of Neuroma | 2 years
  Recurrence of neuroma as assessed by clinical assessment by the surgeon.
Elliot Neuroma questionnaire | 2 years
  Type of pain
QuickDASH | 2 years
  Daily functioning upper limb
Goals questionnaire | 2 years
  Daily functioning lower limb
Type of Pain Medication | 2 years
  Type of pain medication currently taken
Amount of Pain Medication | 2 years
  Amount of pain medication currently taken

CONTACTS AND LOCATIONS:
Locations (16):
- United States (8):
  - Arizona Center for Hand Surgery, Phoenix, Arizona
  - Stanford Medical Center Hand and Upper Limb Center, Redwood City, California
  - Buncke Clinic, San Francisco, California
  - Veterans affairs Medical Center Portland, Portland, Oregon
  - Geisinger Clinic, Danville, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The Philadelphia Hand Center (affiliated to Thomas Jefferson Hospital), Philadelphia, Pennsylvania
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
- Clinique Chirurgicale Victor Hugo Paris, Paris, France
- BG Trauma Center Frankfurt am Main GmbH, Frankfurt am Main, Germany
- Ospedale San Guiseppe Milano, Milan, Italy
- Parc Sanitari Sant Joan de Deu, Barcelona, Spain
- Sweden (3):
  - Sahlgrenska University Hospital Gothenburg, Gothenburg
  - University Hospital Linköping, Linköping
  - University Hospital Lund - Department of Hand Surgery, Malmo
- Birmingham Hand Centre, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Power D, Curtin C, Bellemere P, Nyman E, Pajardi G, Isaacs J, Levin LS. Surgical Treatment of Symptomatic End-Neuroma With a New Bioresorbable Copolyester Nerve Capping Device: A Multicenter Prospective Cohort Study. Ann Plast Surg. 2023 Jul 1;91(1):109-116. doi: 10.1097/SAP.0000000000003596. PMID 37450869